CLINICAL TRIAL: NCT01403376
Title: Study to Investigate the Immune Response to Influenza Vaccine in Patients With Multiple Sclerosis on Teriflunomide Treatment and Using a Population of Patients With Multiple Sclerosis as a Reference
Brief Title: Study to Investigate the Immune Response to Influenza Vaccine in Patients With Multiple Sclerosis on Teriflunomide
Acronym: TERIVA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: PDY11684; 2011-001160-21 (EudraCT Number: UTN); U1111-1115-2742 (Other: UTN)
Record Dates: First submitted 2011-07-14; First posted 2011-07-27 (Estimated); Results first posted 2013-02-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — teriflunomide; Interferon beta-1a; Interferon beta-1b; Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Teriflunomide 7 mg (Experimental): Influenza vaccine in participants treated with teriflunomide 7 mg for at least 6 months
  Interventions: Drug: teriflunomide; Biological: Influenza vaccine
- Teriflunomide 14 mg (Experimental): Influenza vaccine in participants treated with teriflunomide 14 mg for at least 6 months
  Interventions: Drug: teriflunomide; Biological: Influenza vaccine
- IFN-β-1 (Active Comparator): Influenza vaccine in participants treated with a stable dose of Interferon-β-1 (IFN-β-1) for at least 6 months
  Interventions: Drug: Interferon-β-1; Biological: Influenza vaccine

INTERVENTIONS:
Drug: teriflunomide — Film-coated tablet
  Oral administration
  Other Names: HMR1726
  Arms: Teriflunomide 14 mg; Teriflunomide 7 mg
Drug: Interferon-β-1 — Powder for reconstitution, of any licensed strength for either intramuscular or subcutaneous injection
  Other Names: Rebif®; Avonex®; Betaseron®; Betaferon®; Extavia®; Genfaxone®
  Arms: IFN-β-1
Biological: Influenza vaccine — Inactivated, split-virion influenza vaccine 2011-2012
  One administration by intramuscular or intradermal route as per product specification

SUMMARY:
Primary Objective:

Assess the antibody response to influenza vaccine in patients with relapsing form of multiple sclerosis (RMS) treated with teriflunomide compared to a reference population.

Secondary Objectives:

* Assess the effect of teriflunomide on immunoglobulin levels;
* Assess the safety of influenza vaccination in patients with RMS treated with teriflunomide.

The reference population was defined as multiple sclerosis (MS) patients with a stable treatment with interferon-β-1. Antibody response was measured using hemagglutination inhibition assay (HIA) and the hemagglutinin antigens representing the stains of H3N2, H1N1, and B as present in the influenza vaccine used.

DETAILED DESCRIPTION:
The maximum duration of the study period for a participant was approximatively 49 days broken down as follows:

* Screening period of up to 21 days;
* Influenza vaccination at Day 1;
* Follow-up period of 28 days (±2 days).

MS treatment (Teriflunomide or interferon-β-1) was to be continued during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

- Male or female patient <60 years old with relapsing multiple sclerosis (RMS) either treated for at least 6 months with 7 or 14 mg teriflunomide in one of the studies LTS6048 or LTS6050, or treated with a stable dose of interferon-β-1 for at least 6 months.

Exclusion Criteria:

* Concomitant infectious pathology at the time of vaccination;
* MS relapse within 1 month before vaccination;
* Systemic corticosteroids within 1 month before the vaccination;
* Any contraindication to influenza vaccine;
* Any vaccination within the last 6 months;
* Prior use of any investigational drug or participation to a clinical trial within 1 year (only for patients under interferon-β-1);
* Prior or concomitant use (for a minimum of 1 year before study entry) of cladribine, mitoxantrone, or other immunosuppressant agents such as azathioprine, cyclophosphamide, cyclosporin, methotrexate, mycophenolate, natalizumab (Tysabri®), leflunomide or fingolimod or other immunomodulator/immunosuppressant in development;
* Prior or concomitant use of glatiramer acetate within 1 year before study entry;
* Prior or concomitant use of intravenous immunoglobulins within 3 months before study entry;
* Pregnant or breast feeding women;
* Woman of childbearing potential without adequate contraception.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2011-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (14):
- Investigational Site Number 040001, Vienna, Austria
- Canada (7):
  - Investigational Site Number 124005, Calgary
  - Investigational Site Number 124003, Greenfield Park
  - Investigational Site Number 124002, London
  - Investigational Site Number 124007, Montreal
  - Investigational Site Number 124008, Ottawa
  - Investigational Site Number 124001, Québec
  - Investigational Site Number 124009, Toronto
- Germany (3):
  - Investigational Site Number 276003, Berlin
  - Investigational Site Number 276001, Essen
  - Investigational Site Number 276002, Münster
- Investigational Site Number 643002, Nizhny Novgorod, Russia
- Ukraine (2):
  - Investigational Site Number 804002, Ivano-Frankivsk
  - Investigational Site Number 804001, Kharkiv

REFERENCES:
- [Result] Bar-Or A, Freedman MS, Kremenchutzky M, Menguy-Vacheron F, Bauer D, Jodl S, Truffinet P, Benamor M, Chambers S, O'Connor PW. Teriflunomide effect on immune response to influenza vaccine in patients with multiple sclerosis. Neurology. 2013 Aug 6;81(6):552-8. doi: 10.1212/WNL.0b013e31829e6fbf. Epub 2013 Jul 12. PMID 23851964

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment initiated in September 2011 was completed in December 2011. A total of 137 patients were screened at 14 sites in 5 countries.
  Participants treated with teriflunomide were recruited in the LTS6048-NCT00228163 study and in the LTS6050-NCT00803049 study.
Pre-assignment Details: In order to ensure at least 40 participants were enrolled in the teriflunomide 14 mg group while maintaining the blind in the study LTS6050 an interactive voice response system (IVRS) was set up to include participants from both studies LTS6048 and LTS6050 into this study.
  128 participants were enrolled and vaccinated at 14 sites.
Period: Overall Study
Arm/Group | Teriflunomide 7 mg | Teriflunomide 14 mg | IFN-β-1
Started | 41 | 41 | 46
Completed | 41 | 41 | 46
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teriflunomide 7 mg | Teriflunomide 14 mg | IFN-β-1 | Total
Number analyzed (Participants) | 41 | 41 | 46 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (7.9) | 43.8 (8.5) | 45.1 (10.8) | 45.0 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 32 | 89
  Male | 13 | 12 | 14 | 39
pre-vaccination antibody titer - H1N1 strain [Number; unit: participants] — H1N1, H3N2 and B were the strains contained in the seasonal influenza vaccine used.
  participants
    <10 | 0 | 1 | 0 | 1
    Between 10 and 40 (<) | 7 | 4 | 5 | 16
    ≥40 | 34 | 36 | 41 | 111
pre-vaccination antibody titer - H3N2 strain [Number; unit: participants]
  <10 | 2 | 3 | 2 | 7
  Between 10 and 40 (<) | 16 | 15 | 22 | 53
  ≥40 | 23 | 23 | 22 | 68
pre-vaccination antibody titer - B strain [Number; unit: participants]
  <10 | 0 | 0 | 0 | 0
  Between 10 and 40 (<) | 12 | 13 | 21 | 46
  ≥40 | 29 | 28 | 25 | 82

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Antibody Titer ≥40 at 28 Days Post Vaccination
Description: For each viral strain (H1N1, H3N2, and B), the antibody titer, level of antibodies in blood sample when exposed to antigen, was calculated as the mean of two replicates. If the titer was below or above the limit of detection, the threshold value was used.
  The percentage of participants achieving a titer of 40 or more, as well as the 90% confidence interval (CI) using normal approximation were calculated for each strain and treatment group.
Time Frame: 28 days post vaccination
Population: Per-protocol population: Enrolled and vaccinated participants with antibody assessments at Day 28, but excluding those with important events/deviations potentially impacting analysis (multiple sclerosis relapse, poor compliance to treatment, interfering concomitant drug). Participants were considered according to the treatment actually received.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Teriflunomide 7 mg | Teriflunomide 14 mg | IFN-β-1
Number analyzed (Participants) | 40 | 39 | 43
percentage of participants
  H1N1 strain | 97.5 [93.4 to 100.0] | 97.4 [93.3 to 100.0] | 97.7 [93.9 to 100.0]
  H3N2 strain | 90.0 [82.2 to 97.8] | 76.9 [65.8 to 88.0] | 90.7 [83.4 to 98.0]
  B strain | 97.5 [93.4 to 100.0] | 97.4 [93.3 to 100.0] | 93.0 [86.6 to 99.4]

2. Secondary Outcome: Percentage of Participants With 2 Fold or More Increase in Antibody Titer at 28 Days Post Vaccination
Description: Percentages of participants with an increase from baseline of 2-fold or more in antibody titers and 90% CIs using normal approximation were calculated for each strain and treatment group.
Time Frame: pre vaccination (baseline) and 28 days post vaccination
Population: Per-protocol population as previously defined
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Teriflunomide 7 mg | Teriflunomide 14 mg | IFN-β-1
Number analyzed (Participants) | 40 | 39 | 43
percentage of participants
  H1N1 strain | 35.0 [22.6 to 47.4] | 30.8 [18.6 to 42.9] | 46.5 [34.0 to 59.0]
  H3N2 strain | 35.0 [22.6 to 47.4] | 41.0 [28.1 to 54.0] | 51.2 [38.6 to 63.7]
  B strain | 47.5 [34.5 to 60.5] | 51.3 [38.1 to 64.4] | 58.1 [45.8 to 70.5]

3. Secondary Outcome: Percentage of Participants With 4 Fold or More Increase in Antibody Titer at 28 Days Post Vaccination
Description: Percentages of participants with an increase from baseline of 4-fold or more in antibody titers and 90% CIs using normal approximation were calculated for each strain and treatment group.
Time Frame: pre vaccination (baseline) and 28 days post vaccination
Population: Per-protocol population as previously defined
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Teriflunomide 7 mg | Teriflunomide 14 mg | IFN-β-1
Number analyzed (Participants) | 40 | 39 | 43
percentage of participants
  H1N1 strain | 22.5 [11.6 to 33.4] | 20.5 [9.9 to 31.1] | 39.5 [27.3 to 51.8]
  H3N2 strain | 25.0 [13.7 to 36.3] | 23.1 [12.0 to 34.2] | 41.9 [29.5 to 54.2]
  B strain | 37.5 [24.9 to 50.1] | 30.8 [18.6 to 42.9] | 51.2 [38.6 to 63.7]

4. Secondary Outcome: Geometric Mean of Titers (GMT) Ratio Post/Pre Vaccination
Time Frame: pre vaccination (baseline) and 28 days post vaccination
Population: Per-protocol population as previously defined
Measure: Geometric Mean (90% Confidence Interval); unit: ratio post/pre vaccination
Arm/Group | Teriflunomide 7 mg | Teriflunomide 14 mg | IFN-β-1
Number analyzed (Participants) | 40 | 39 | 43
ratio post/pre vaccination
  H1N1 strain | 2.5 [2.0 to 3.3] | 2.3 [1.9 to 2.9] | 3.4 [2.6 to 4.5]
  H3N2 strain | 2.6 [1.9 to 3.5] | 2.6 [1.9 to 3.6] | 4.1 [3.0 to 5.4]
  B strain | 3.1 [2.3 to 4.2] | 3.0 [2.3 to 3.9] | 4.7 [3.6 to 6.2]

5. Secondary Outcome: Immunoglobulin Levels
Time Frame: pre vaccination (baseline) and 28 days post vaccination
Population: Per-protocol population as previously defined
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Teriflunomide 7 mg | Teriflunomide 14 mg | IFN-β-1
Number analyzed (Participants) | 40 | 39 | 43
g/L
  Immunoglobulin M - pre vaccination | 1.28 (0.57) | 1.23 (0.59) | 1.14 (0.58)
  Immunoglobulin M - 28-day post vaccination | 1.30 (0.56) | 1.27 (0.60) | 1.16 (0.54)
  Immunoglobulin G - pre vaccination | 9.35 (1.82) | 9.12 (2.24) | 12.03 (3.01)
  Immunoglobulin G - 28-day post vaccination | 9.57 (2.08) | 9.09 (2.25) | 12.25 (2.69)
  Immunoglobulin A - pre vaccination | 1.65 (0.66) | 1.51 (0.64) | 2.27 (1.07)
  Immunoglobulin A - 28-day post vaccination | 1.63 (0.68) | 1.50 (0.63) | 2.33 (1.07)

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected from signature of the Informed Consent Form (ICF) up to the last visit in the study.
Description: The analysis was performed on the included and vaccinated population and included all AE that developed or worsened from vaccination up to the end of study visit at Day 28.
Groups:
- Teriflunomide 7mg: Influenza vaccine in participants treated with teriflunomide 7 mg for at least 6 months
- Teriflunomide 14mg: Influenza vaccine in participants treated with teriflunomide 14 mg for at least 6 months
Arm/Group | Teriflunomide 7mg | Teriflunomide 14mg | IFN-β-1
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41 | 0/46
Other Adverse Events (participants affected / at risk) | 3/41 | 6/41 | 13/46
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Teriflunomide 7mg (N=41) | Teriflunomide 14mg (N=41) | IFN-β-1 (N=46)
Nasopharyngitis (Infections and infestations) | 2 | 3 | 6
Headache (Nervous system disorders) | 1 | 1 | 3
Influenza like illness (General disorders) | 0 | 1 | 4
Injection site pain (General disorders) | 1 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months after trial completion, the Investigator can present or publish results. The Investigator provides the Sponsor with a copy of the presentation or publication for review and comment at least 30 days in advance of its submission.

The Sponsor can delay the submission for a period not exceeding 90 days to allow for filing a patent application or such other measures as the Sponsor deems appropriate to establish and preserve its proprietary rights.